CLINICAL TRIAL: NCT06586203
Title: New GENOmic Predictor for COmplications Risk in Type 2 DIAbetes
Brief Title: Clinical Utility of a Genomic Predictor Test on the Management of Cardiorenal Complications of Type 2 Diabetes
Acronym: GENOCORDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optithera (Industry)
Collaborators: Genome Quebec (Other); Genome Canada (Other); ELNA Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPT0003
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetic Nephropathy Type 2
Keywords: Diabetes Mellitus, Type 2; Cardiorenal complications; Polygenic risk scores; Therapeutic targets; Precision Medicine; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Genetic Risk Score

STUDY DESIGN:
Intervention Model Description: A) A pragmatic trial designed to evaluate the effectiveness of GENOCORDIA PRS testing in real-life routine practice conditions.
  B) Randomization of participants into informed and uninformed populations of the Polygenic risk score test result.
  C) Adaptive trial for the treatment of subjects initially uninformed of their PRS test result after 12 months if positive results.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informed (Active Comparator): Intervention group tested and informed of the Polygenic risk score test result at the start of the study
  Interventions: Device: Polygenic Risk Score
- Not initially informed (No Intervention): Control group: tested but not informed of the Polygenic Risk Score test result at the start of the study.

INTERVENTIONS:
Device: Polygenic Risk Score — The Polygenic Risk Score (PRS) is a Class II software as a medical device (SaMD) that estimates a person's level of risk of developing a disease or associated complications before clinical signs appear. The device uses the genomic profile of the person in combination with some clinical data (i.e., age, sex, age of onset of diabetes) to compute this risk. This device further provides recommendations for personalized management of T2D for patients based on their risk score.
  Other Names: Risk Prediction
  Arms: Informed

SUMMARY:
The goal of this pragmatic trial is to provide Real World Evidence (RWE) on the impact of the result of a polygenic risk prediction test of cardiorenal complications of T2D, so that more patients at high risk of these complications achieve over an 18 months period, recommended therapeutic targets.

This will be demonstrated as a significant improvement in a composite value including HbA1c or systolic blood pressure (SBP) or albuminuria (UACR), or glomerular filtration rate (GFR) lowering.

Researchers will compare the recommended therapeutic targets of uninformed and informed patients to see if the knowledge of the risk by the patients and their treating physicians improves achievement of these targets.

Participants will:

Have a saliva sampling to determine the genetic risk. Visit the clinic once every 3 months for checkups and tests Answer two questionnaires on quality of life.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) increases the risk of developing serious cardiovascular and kidney complications that represent a major burden for both patients and our healthcare system. Currently, patients with T2D are treated according to guidelines, with varied results in terms of systolic blood pressure (SBP), blood glucose (HbA1c), urine albumin-creatinine ratio (UACR) and glomerular filtration rate (GFR) target achievement.

OPTITHERA has developed the first genomic test to predict the risk of cardiorenal complications that will allow early and personalized treatment of patients with T2D who are at high risk using Polygenic risk score.

It is proposed that knowledge of the risk of developing complications of diabetes will have a positive effect on the care pathway of diabetic patients: the patient will be able to actively participate in their care and their doctor will be able to adapt his treatment to his personal risk, especially if his patient is at high risk of complications.

Objective: To provide Real World Evidence (RWE) on the impact of the result of a PRS prediction test on the risk of complications of T2D, so that patients at high risk of complications achieve, over an 18-month period, recommended targets for systolic blood pressure (≤130 mmHg) or HbA1c (<7.0%), or decreased albuminuria grade, GFR decline, while avoiding severe hypoglycemia and falls.

This will be demonstrated as a significant improvement in composite value including HbA1c or systolic blood pressure (SBP) or albuminuria (UACR).

Methodology: Multicenter Study: A) Pragmatic trial designed to evaluate the effectiveness of GENOCORDIA PRS testing in real-life routine practice conditions.

B) Randomization of participants into informed and uninformed populations of the PRS test result. C) Adaptive trial for the treatment of subjects initially uninformed of their PRS test result.

Estimated number of participants: 2714 participants randomized into two groups. Estimated study enrollment duration= 9 months. Estimated total study duration = 36 months. 18 months follow-up (7 visits).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with T2D of both sexes regardless of ethnicity, level of diabetes control and presence of complications.
* Able to visit the study site 7 times
* Able and willing to provide informed consent to the clinical and PRS parts of the study.

Exclusion Criteria:

* Any condition that may impact participation in a real-world study according to the treating physician.
* People with a high frailty index as no benefit of therapeutic intensification has been demonstrated in these diabetic patients.
* People who refuse to be informed of their cardiorenal risk score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2714 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2028-08-23 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint consisting of HbA1c, SBP, albuminuria or GFR | Visit to visit up to 18 months
  Change of HbA1c, or SBP or albuminuria stage or eGFR decline. Percent of participants at therapeutic targets.

SECONDARY OUTCOMES:
Medications for blood pressure, blood glucose and lipids | Visit to vist up to 18 months
  change of class or dosage

OTHER OUTCOMES:
Microvascular and macrovascular endpoints | 18 months
  Macrovascular outcome comprises nonfatal stroke, nonfatal acute coronary syndrome and death from any cardiovascular cause. Microvascular endpoint comprises new or worsening nephropathy defined as the development of macroalbuminuria, doubling of serum creatinine, requirement for renal replacement therapy or death from renal disease.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Hamet, MD, PhD, Principal Investigator — CHUM
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - ELNA Medical, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data at the end of the study including risk strata.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Six months after study publication.
Access Criteria: Contact the PI.

REFERENCES:
- [Background] Tremblay J, Haloui M, Attaoua R, Tahir R, Hishmih C, Harvey F, Marois-Blanchet FC, Long C, Simon P, Santucci L, Hizel C, Chalmers J, Marre M, Harrap S, Cifkova R, Krajcoviechova A, Matthews DR, Williams B, Poulter N, Zoungas S, Colagiuri S, Mancia G, Grobbee DE, Rodgers A, Liu L, Agbessi M, Bruat V, Fave MJ, Harwood MP, Awadalla P, Woodward M, Hussin JG, Hamet P. Polygenic risk scores predict diabetes complications and their response to intensive blood pressure and glucose control. Diabetologia. 2021 Sep;64(9):2012-2025. doi: 10.1007/s00125-021-05491-7. Epub 2021 Jul 6. PMID 34226943